CLINICAL TRIAL: NCT05042817
Title: Effect of Intrathecal Morphine on Urinary Bladder Function and Recovery in Patients Having a Cesarean Delivery - A Double-blind Randomized Clinical Trial
Brief Title: Effect of Intrathecal Morphine on Urinary Bladder Function and Recovery in Patients Having a Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean François Brichant, Principal investigator, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VesicalMorphine
Record Dates: First submitted 2021-08-16; First posted 2021-09-13 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Analgesia
Keywords: Obstretics; Regional anesthesia; Injections; Spinal; Analgesics; Opioid
MeSH Terms: conditions — Agnosia | interventions — Morphine; Saline Solution; Prilocaine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patient assessments and bladder urodynamic data collection were performed by two blinded anesthesiologists.
  Randomization was performed using the sealed envelopes method. Therefore, one of the anesthesiologists of the research team, who was unblinded, opened the envelopes and prepared the injection mixtures.
  Another two blinded anesthesiologists administered perioperative anesthesia and monitored the patient during the perioperative period, and evaluated sensitive and motor block.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morphine (Active Comparator): 50 mg prilocaine + 2.5 mcg sufentanil + 100 mcg morphine (0.1ml)
  Interventions: Drug: 100 mcg morphine; Drug: 50 mg prilocaine + 2.5 mcg sufentanil
- NaCl 0.9% (Placebo Comparator): 50 mg prilocaine + 2.5 mcg sufentanil + 0.1 ml saline
  Interventions: Drug: 0.9% NaCl; Drug: 50 mg prilocaine + 2.5 mcg sufentanil; Procedure: bilateral transverse abdominal plane block

INTERVENTIONS:
Drug: 100 mcg morphine — The effect of intrathecal morphine on vesical function and the need for bladder re-catheterization after a cesarean delivery
  Arms: Morphine
Drug: 0.9% NaCl — NaCl 0.9%
  Arms: NaCl 0.9%
Drug: 50 mg prilocaine + 2.5 mcg sufentanil — 50 mg prilocaine + 2.5 mcg sufentanil
Procedure: bilateral transverse abdominal plane block — 20 mL of ropicavaine 0.375% on each side
  Other Names: TAP block
  Arms: NaCl 0.9%

SUMMARY:
The enhanced recovery anesthesia concept has been widely adopted, including cesarean delivery. Modern obstetrical anesthesia aims to offer an experience to a patient undergoing a cesarean delivery similar to normal vaginal delivery in order to maximize postoperative comfort and facilitate bonding between the mother and her newborn. Therefore, early removal of the bladder catheter has been recommended. However, this is challenged by the administration of intrathecal morphine recommended to provide long-lasting postoperative analgesia after cesarean delivery.

DETAILED DESCRIPTION:
This double-blind, randomized trial investigates the effects of intrathecal morphine on urinary dynamics in women undergoing CD under spinal anesthesia. The hypothesis is that the addition of intrathecal morphine (ITM) will delay micturition in women undergoing cesarean delivery. The primary outcome is the effect of ITM on urodynamics the difference in time to micturition. The secondary outcome is the need for bladder re-catheterization.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I and II
* Term singleton pregnancies
* Elective cesarean delivery under spinal anesthesia
* Between October 2021 and March 2022

Exclusion Criteria:

* Pre-existing or gestational hypertension
* Diabetes
* Cardiovascular disease
* Cerebrovascular disease
* Known fetal abnormalities
* Extremes of weight (<40 kg or > 100 kg)
* Contraindications to neuraxial anesthesia
* Twin pregnancies
* Excessive intraoperative bleeding (blood loss exceeding > 1000 mL or requiring a blood transfusion)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women with term singleton pregnancies are included, therefore males cannot be included
Enrollment: 56 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
First micturition (hours) | until the end of the study, an average of 6 months
  Vesicle function 1
Bladder volume (mL) | until the end of the study, an average of 6 months
  Vesicle function 2
Debimetry | until the end of the study, an average of 6 months
  Vesicle function 3

SECONDARY OUTCOMES:
Bladder re-catherization | until the end of the study, an average of 6 months
  Vesicle function 4

CONTACTS AND LOCATIONS:
Locations (1):
- University of Liege, University Hospital, Liège, Belgium